CLINICAL TRIAL: NCT05836805
Title: A Phase 1,Single-center,Open-label Study Investigating the Mass Balance,Pharmacokinetics and Metabolism of [14C]XZP-3621 in Healthy Male Subjects
Brief Title: A Study of the Absorption, Metabolism and Excretion of [14C]XZP-3621 in Human
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XZP-3621-1004
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: [14C]XZP-3621; Mass Balance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]XZP-3621 (Experimental): Eligible healthy 6 volunteers will receive a single oral dose of 400 mg/200 µCi [14C]XZP-3621 administered by mouth, as a suspension solution.
  Interventions: Drug: [14C]XZP-3621

INTERVENTIONS:
Drug: [14C]XZP-3621 — Extemporaneously compounded oral suspension solution of [14C]XZP-3621 (400 mg/200 µCi)

SUMMARY:
This non-randomized, single group, open-label study will investigate the mass balance, routes of elimination, pharmacokinetics, metabolism, safety and tolerability of a single oral dose of [14C]XZP-3621 in healthy volunteers.

DETAILED DESCRIPTION:
This open-label, radiolabeled, single 400-mg dose study in approximately 6 healthy male volunteers has been designed to further the understanding of human metabolism of XZP-3621.

Subjects who had signed informed consent and meet inclusion criteria and no exclusion criteria are admitted to Phase I Clinical Unit two days prior to dosing (D-2). On the morning of Day 1 before dosing, subjects will be performed baseline examination and trained on procedures such as medicine-taking, PK blood collection, urine and fecal collection, etc., to ensure that the procedures can be performed according to the protocols and standard operating procedures. And after an overnight fast of at least 10 h, 30 minutes afer a standard meal, subjects will receive a single oral dose of 400 mg (200 μCi) of [14C]XZP-3621 as an oral suspension. Water will be banned from 1 hour pre-dose to 1 hour post-dose (excluding when taking the medicine) and food will be banned within 4 hours post-dose.

Metabolic profiling of radiolabeled components will be performed on pooled plasma samples as well as on cumulative urine and feces excreted until Day 14 postdose or until one of the early release criteria is met. The early release criteria are: 1) recovery in excreta of at least 80% of administered radioactivity, or 2) less than 1% of administered radioactivity being recovered in excreta from two consecutive days (ie, total for urine + feces should be <1% on 2 consecutive days).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

A subject will be eligible for study participation if he meets the following criteria:

1. healthy male volunteers between the ages of 18 to 45 years old, inclusive 18 and 45;
2. Body weight >=50 kg, Body mass index (body weight(kg)/hight2(m2)) between 19 and 26 kg/m2 (inclusive);
3. Male subjects of reproductive potential with partners will be instructed to, and must be willing to practice a highly effective method of birth control for the duration of the study and continuing 1 year after discontinuing treatment with the investigational product. Highly effective methods of birth control include using condom, contraceptive sponge, contraceptive gel, contraceptive film, intrauterine device, oral or injectable contraceptive pill, hypodermic implants or others;
4. Must understand, and voluntarily sign the informed consent, comply with the requirements of the study.

Exclusion Criteria:

* A subject will not be eligible for study participation if he meets any of the exclusion criteria:

  1. Allergies, have allergies to two or more drugs or foods; or have known allergies to the components of the test drug;
  2. Clinically significant medical history or findings in physical examination, vital signs, or laboratory test results prior to study start;
  3. Clinically significant of ophthalmologic examinations;
  4. Positive test for HBsAg, HBeAg, anti-HCV, anti-HIV or syphilis antibody;
  5. History of or current swallowing disorder, active gastrointestinal diseases, or other diseases that significantly affect absorption, distribution, metabolism and excretion of drugs;
  6. History of or current clinically significant cardio, pulmonary, endocrine, metabolism, renal, hepatic, gastrointestinal, dermatology, infection, hematology, neurological, mental disease or disorder;
  7. Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease,Hemorrhoids or perianal disease with regular/perianal bleeding;
  8. Received major surgery within 6 months prior to the screening period or surgical incisions were not fully healed;
  9. Smoking (> 5 cigarette / day), drinking (> 14 units, pure alcohol / week, equivalent to 360 ml beer/unit, or 45 ml low-alcohol liquor) within 3 months prior to the screening period or Positive screening tests for alcohol,Subjects should avoid smoking and drinking during the clinical trail;
  10. Participation in an investigational drug or device study within 3 months prior to screening period;
  11. Subjects who have participated in radiolabeled clinical study within 1 year prior to screening period;
  12. History of abusing drugs(MOP, METmAMP, MTD, THC, AMP positive) within 1 year prior to screening period;
  13. Have donated 400ml or more of blood or plasma 3 months prior to the study drug administration;
  14. Received any drug within 14 days before taking the investigational drug, including any prescription drug, OTC drug or herbal drug;
  15. Use of any metabolic inducers (including herbals such as St. John's Wort) or inhibitors within 14 days before the first dose of study medication;
  16. Failure to comply with clinical study protocols, such as non-cooperation, follow-up visit and completion of entire study;
  17. Vaccination was administered within 1 months prior to screening or during screening;
  18. Significant radiation exposure within one year prior to drug administration (more than 2 exposures from chest X-ray or CT scan, or barium meal examination and radiation-related occupations);
  19. Investigators think that subjects are not suitable to participate in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Total recovery of radioactivity in urine and feces | Assessments will be made up to 19 days post dose
  Calculate the total radioactivity in urine and feces based on the radioactivity concentration of each sample.
Radioactivity concentration of each plasma sample | Assessments will be made up to 19 days post dose
  Use liquid scintillation counter to evaluate Radioactivity concentration of each plasma(DPM/ml) sample
Metabolic profiling for XZP-3621 will be determined in plasma, urine and fecal samples | Assessments will be made up to 19 days post dose
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in plasma, urine and feces.
Maximum exposure in plasma will be determined for XZP-3621, XZP-5089 metabolite and total radioactivity | Assessments will be made up to 19 days post dose
  Cmax (maximum observed plasma concentration) will be reported directly from each analyte's data
The overall exposure in plasma will be determined for XZP-3621, metabolite and total radioactivity | Assessments will be made up to 19 days post dose
  AUC0-∞ (Area under the plasma concentration time profile from time 0 extrapolated to infinite time) will be determined, using Linear/Log trapezoidal method, from plasma concentration data for each analyte
The terminal elimination half life in plasma will be estimated from plasma profiles over time for XZP-3621, metabolite and total radioactivity | Assessments will be made up to 19 days post dose
  t1/2 (apparent terminal elimination half life) will be estimated for each analyte from the terminal portion of its plasma concentration versus time plot

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Assessments will be made up to 28 days post dose
  According to CTCAE v5.0, the number and frequency of adverse events after a single dose of [14C]XZP-3621 were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, DPH, Principal Investigator — First Affiliated Hospital of Suzhou Medical College
Locations (1):
- The First Affiliated Hospital of Suzhou Universiy, Suzhou, Jiangsu, China